CLINICAL TRIAL: NCT06543797
Title: A Prospective, Single-center, Single-group, Investigator-led Exploratory Clinical Trial to Determine the Safety of the Application of a Wearable Medical Electromagnetic Generator.
Brief Title: A Pilot Clinical Trial Study to Determine the Safety of the Application of a Wearable Medical Electromagnetic Generator
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, MD, PhD, Principle investigator, Bundang CHA Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-01-070
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stroke patients (Experimental)
  Interventions: Device: wearable rTMS

INTERVENTIONS:
Device: wearable rTMS — Application of inhibitory low-frequency rTMS on unaffected primary motor cortex by wearable rTMS

SUMMARY:
To explore the safety of applying repetitive low-frequency transcranial magnetic stimulation using a wearable medical electromagnetic generator in stroke patients.

ELIGIBILITY:
Inclusion criteria

1. Patients aged 19 to 80 years old
2. Those who are confirmed to have lesions in only one cerebral hemisphere or one brainstem on brain computed tomography (CT) or brain magnetic resonance imaging (MRI)
3. Patients with subacute stroke between 2 weeks and less than 3 months after onset
4. Motor function evaluation The total score is 0 to 56 points based on the FMA of the upper extremity on the affected side [1], and patients show impairment in upper extremity motor function.
5. After receiving a detailed explanation of this clinical trial and fully understanding it, the subject or legal representative voluntarily decides to participate and agrees in writing to comply with the precautions.

Exclusion Criteria:

1. Cases accompanied by existing serious neurogenic diseases such as history of underlying stroke, brain tumor, hypoxic brain injury, epilepsy, or organic brain disease
2. Cases accompanied by existing serious psychiatric diseases such as major schizophrenia, bipolar disorder, dementia, etc., that are receiving continuous drug treatment before the stroke.
3. Those with unstable conditions in the cardiovascular, digestive, respiratory, and endocrine systems, or with severe internal diseases such as signs of systemic infection, with unstable vital signs, or with poor overall health with a life expectancy of less than 1 year.
4. Those with impaired cognitive ability (MMSE less than 10 points)
5. If there are difficulties in conducting research
6. If you have difficulty communicating
7. Other patients who are deemed difficult to participate in this study by the principal investigator.
8. Patients who are participating in other therapeutic clinical studies or who have participated in other therapeutic clinical studies within the past 30 days (observational studies are not relevant)
9. Exclusion criteria for repetitive transcranial magnetic stimulation
10. Patients with medical devices implanted in the body (e.g. pacemaker)
11. When a metal object is inserted into the skull
12. If there is a wound on the skin at the attachment site
13. History of epilepsy
14. If you have cervical pain or musculoskeletal disease
15. Pregnant and lactating women

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety | Before and after 2 weeks of intervention / Soon after every intervention
  All types of adverse events that occurred during clinical trials

SECONDARY OUTCOMES:
Changes of Fugl-Meyer assessment | Before and after 2 weeks of intervention
  Fugl-Meyer assessment for motor function in score
Changes of manual muscle test (MMT) | Before and after 2 weeks of intervention
  Manual muscle test for strength in score
Changes of box and block test (BBT) | Before and after 2 weeks of intervention
  Box and block test for gross manual dexterity in number of blocks from on compartment of a box to another of equal size within 60 seconds
Changes of action research arm test (ARAT) | Before and after 2 weeks of intervention
  Action research arm test for functional ability of upper extremity in score
Changes of Korean mini-mental state examination (K-MMSE) | Before and after 2 weeks of intervention
  Korean mini mental state exam for cognitive function in score
Changes of Korean version of Modified Barthel Index (K-MBI) | Before and after 2 weeks of intervention
  Korean version of modified barthel index for functional status in score
Changes of geriatric depression scale (GDS-d) | Before and after 2 weeks of intervention
  Geriatric depression scale for depression in scale
Changes of electroencephalograpy (EEG) | Before and after 2 weeks of intervention
  Electroenchphalography is a test that measures EEG power in alpha band
Changes of Evoked-potentials (EP) | Before and after 2 weeks of intervention
  Evoked potential is an electrical potential recorded from the nervous system of a human or animal following presentation of a stimulus. In this study, motor- and sensory- evoked potentials are included.
Changes of motion analysis | Before and after 2 weeks of intervention
  Motion analysis with motion capture setup and data processing or streaming of patients movements. In this study, data of motion capture include kinetic and kinematic data including physiological parameter.
Changes of functional near-infrared spectroscopy (fNIRS) | Before and after 2 weeks of intervention
  Funtional near-infrared spectroscopy meausures cortical activity in concentration of oxy- and deoxy-hemoglobin
Changes of blood biomarker | Before and after 2 weeks of intervention
  Blood biomarker include expression of tumor necrosis factor (TNF)-a and interleukin (IL)-1b

CONTACTS AND LOCATIONS:
Overall Officials: Minyoung Kim, M.D., Ph.D., Principal Investigator — Bundang CHA Hospital

IPD SHARING:
Plan to Share IPD: No